CLINICAL TRIAL: NCT07240974
Title: A Clinical Study to Evaluate the Safety and Efficacy of ZZSW-01 in the Treatment of Patients With Relapsed/Refractory B-cell Malignancies
Brief Title: Safety and Efficacy of ZZSW-01 in Relapsed/Refractory B-cell Malignancies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, MEI HENG, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVB20250627
Record Dates: First submitted 2025-09-03; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Relapsed/Refractory B-cell Malignancies
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZZSW-01 (Experimental): ZZSW-01 is an extracellular vesicle that carries functional CD19 CAR mRNA, which can be administered intravenously to generate CAR-T cells in vivo.
  Interventions: Drug: ZZSW-01 injection

INTERVENTIONS:
Drug: ZZSW-01 injection — ZZSW-01 is an extracellular vesicle that carries functional CD19 CAR mRNA, which can be administered intravenously to generate CAR-T cells in vivo.
  Other Names: CAR-EVs

SUMMARY:
This is a single-center, single-arm, open-label, dose-escalation, early-phase 1 study to evaluate the safety, tolerability and preliminary efficacy of ZZSW-01 injection in patients with relapsed/refractory B-cell malignancies.

DETAILED DESCRIPTION:
This investigator-initiated clinical study aims to evaluate ZZSW-01 injection, the extracellular vesicle vector that carries CD19 CAR mRNA, in patients with relapsed/refractory B-cell hematologic malignancies. Under this design, eligible subjects will receive multiple injections. The study adopts a dose-escalation design to assess safety, tolerability, and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria:

1. Age ≥18 years, no restriction on sex.
2. ECOG (Eastern Cooperative Oncology Group) performance status score of 0-2.
3. Expected survival ≥3 months.
4. Histologically or cytologically confirmed CD19-positive relapsed or refractory B-cell malignancies according to the WHO classification of lymphoid neoplasms, including:

   Relapsed/refractory B-NHL: patients who have failed at least two prior lines of therapy, are intolerant to the toxicity of second-line regimens, or are not eligible for autologous stem cell transplantation, including but not limited to diffuse large B-cell lymphoma (DLBCL) not otherwise specified, DLBCL/high-grade B-cell lymphoma with MYC and BCL2 rearrangements, high-grade B-cell lymphoma not otherwise specified, primary mediastinal B-cell lymphoma, mantle cell lymphoma, grade 3b follicular lymphoma, and transformed large B-cell lymphoma from indolent B-NHL.

   Relapsed/refractory precursor B-ALL: patients who relapse after achieving CR following second-line therapy, or who fail to achieve CR/CRi after completion of second-line therapy.
5. For relapsed/refractory B-NHL: at least one measurable lesion as assessed by the investigator (e.g., lymph node with long axis >15 mm, or extranodal lesion with long axis >10 mm).

   For relapsed/refractory precursor B-ALL: baseline bone marrow blasts ≥5%.
6. Adequate organ function as defined below (no administration of blood components or hematopoietic growth factors within 14 days prior to first dosing):

   Hematology:

   Relapsed/refractory B-NHL: ANC ≥1.5×10^9/L, platelets ≥75×10^9/L, hemoglobin ≥70 g/L, absolute CD8+ T-cell count ≥0.3×10^9/L; if bone marrow involvement is present: ANC ≥1.0×10^9/L, platelets ≥50×10^9/L, hemoglobin ≥70 g/L.

   Relapsed/refractory precursor B-ALL: ANC ≥1.0×10^9/L (G-CSF support permitted), platelets ≥50×10^9/L (no platelet transfusion within 7 days), hemoglobin ≥80 g/L (no RBC transfusion within 7 days); if bone marrow involvement or not in remission: ANC ≥0.5×10^9/L (G-CSF support permitted), platelets ≥30×10^9/L (no platelet transfusion within 7 days), hemoglobin ≥70 g/L (no RBC transfusion within 7 days). Additionally, absolute CD8+ T-cell count ≥0.2×10^9/L and CD19+ B-cell percentage ≤5%.

   Liver function: TBIL ≤1.5×ULN; ALT and AST ≤2.5×ULN (≤5×ULN if liver metastases are present).

   Renal function: Serum creatinine ≤1.5×ULN (if >1.5×ULN, creatinine clearance must be ≥50 mL/min).

   Coagulation: INR ≤1.5×ULN and APTT ≤1.5×ULN; patients on anticoagulation may be included if INR ≤2.5×ULN.

   Oxygenation: Oxygen saturation >92% on room air.
7. Non-hematologic toxicities from prior therapies (except disease-related) have resolved to ≤grade 1 before enrollment (excluding alopecia and ≤grade 2 neurotoxicity from chemotherapy).
8. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to ZZSW-01 infusion. All fertile male and female participants must agree to use effective contraception during the study and for at least 6 months after the last dose. (Definition of women of childbearing potential and contraceptive methods are detailed in Appendix 1.)
9. Ability and willingness to provide written informed consent and to comply with study procedures, follow-up assessments, and treatment.

Exclusion Criteria

Participants meeting any of the following conditions will be excluded from this study:

1. Patients with CNS involvement of B-cell malignancies confirmed by lumbar puncture and/or MRI with CNS-related symptoms.
2. Patients with isolated extramedullary relapse of B-ALL.
3. Patients with severe hereditary diseases or congenital hematopoietic dysfunction.
4. Patients with Burkitt's lymphoma/leukemia or blast phase chronic myeloid leukemia (p210 BCR-ABL+).
5. Current or past history of central nervous system disorders, including: seizures, ischemic/hemorrhagic cerebrovascular disease, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychiatric illness, or any autoimmune disease involving the CNS.
6. Receipt of chemotherapy within 2 weeks prior to ZZSW-01 infusion (except intrathecal chemotherapy for prevention of CNS leukemia, which must be stopped ≥1 week prior to infusion).
7. Prior systemic immune checkpoint inhibitor therapy (e.g., anti-PD-1/PD-L1 mAbs) within fewer than 3 half-lives before ZZSW-01 infusion; or other systemic antitumor therapy within fewer than 2 weeks or 5 half-lives (whichever is shorter) before infusion.
8. Use of systemic therapeutic corticosteroids within 72 hours prior to ZZSW-01 infusion (physiologic replacement doses are allowed, e.g., prednisone <10 mg/day or equivalent).
9. Receipt of targeted therapies or antibody drugs (including BiTEs, antibody-drug conjugates) within 2 weeks, or cytotoxic therapy within 1 week prior to ZZSW-01 infusion.
10. Autologous stem cell transplantation (ASCT) within 6 weeks prior to ZZSW-01 infusion.
11. Any prior allogeneic hematopoietic stem cell transplantation (allo-HSCT).
12. Known history of the following diseases:

    1. . Systemic vasculitis (e.g., Wegener's granulomatosis, polyarteritis nodosa)
    2. Systemic lupus erythematosus (SLE)
    3. . Active or uncontrolled autoimmune diseases (e.g., Crohn's disease, rheumatoid arthritis, autoimmune hemolytic anemia)
    4. . Primary or secondary immunodeficiency (e.g., HIV infection or severe infectious diseases)
13. Evidence of any of the following infections:

    1. . Chronic or active hepatitis B (HBV) infection (except HBcAb-positive with HBV DNA <500 IU/mL)
    2. . Hepatitis C virus (HCV) infection
    3. . Human immunodeficiency virus (HIV) infection
    4. . Syphilis infection
14. Major surgery within 4 weeks prior to screening, if deemed unsuitable for enrollment by the investigator.
15. Concurrent active malignancy. (Patients with prior malignancies cured ≥2 years may be eligible).
16. Any of the following cardiac conditions:

    1. . Left ventricular ejection fraction (LVEF) ≤45% (by echocardiography)
    2. . NYHA class III or IV congestive heart failure
    3. . Severe arrhythmia requiring treatment, including QTc ≥450 ms in males or ≥470 ms in females (QTcB=QT/RR1/2)
    4. . Uncontrolled hypertension (systolic ≥140 mmHg and/or diastolic ≥90 mmHg), pulmonary hypertension, or unstable angina
    5. . Myocardial infarction, bypass surgery, or stent placement within 12 months prior to dosing
    6. . Clinically significant valvular heart disease
    7. . Any other cardiac disease deemed unsuitable by the investigator
17. Lymphoma involving the atrium or ventricle.
18. Clinical emergencies caused by obstruction or compression from lymphoma masses at screening (e.g., bowel obstruction, vascular compression).
19. History of deep vein thrombosis or pulmonary embolism within 6 months prior to screening.
20. Hypersensitivity (allergy to ≥2 drugs or foods), or known hypersensitivity to components of the investigational product (compound electrolyte injection, 5% human serum albumin).
21. Receipt of live vaccines within 6 weeks prior to screening.
22. Uncontrolled active infection at screening (e.g., sepsis, bacteremia, fungemia, viremia).
23. Participation in another interventional clinical trial with investigational drugs within 3 months prior to ZZSW-01 infusion, or intent to participate in another clinical trial or receive non-protocol antitumor therapy during the study.
24. Any other condition that, in the judgment of the investigator, renders the patient unsuitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Up to 28 days post-infusion
  All adverse events (AEs), including severe adverse events (SAEs) and clinically significant laboratory abnormalities, will be recorded and graded for severity using the Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.
Incidence of Dose-Limiting Toxicities (DLTs) | Up to 28 days post-infusion
  Dose-limiting toxicities (DLTs) will be specifically identified, recorded, and monitored during the designated DLT observation period.
Incidence and Severity of Cytokine Release Syndrome (CRS) | Up to 28 days post-infusion
  Cytokine release syndrome (CRS) events will be identified and graded for severity according to the American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading.
Incidence and Severity of Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) | Up to 28 days post-infusion
  Immune effector cell-associated neurotoxicity syndrome (ICANS) will be assessed using the Immune Effector Cell-Associated Encephalopathy (ICE) score and subsequently graded for severity according to the ASTCT consensus grading.

SECONDARY OUTCOMES:
Complete Response (CR) Rate of administering ZZSW-01 in the treatment of relapsed/refractory of B-cell malignancies. | From ZZSW-01 infusion to the end of the treatment at 96 weeks
  Tumor response after ZZSW-01 infusion will be assessed according to the Lugano 2014 criteria or the 2017 ELN criteria, including complete response (CR).
Partial Response (PR) Rate of administering ZZSW-01 in the treatment of relapsed/refractory of B-cell malignancies. | From ZZSW-01 infusion to the end of the treatment at 96 weeks
  Tumor response after ZZSW-01 infusion will be assessed according to the Lugano 2014 criteria or the 2017 ELN criteria. The Partial Response (PR) rate will be determined.
Stable Disease (SD) Rate of administering ZZSW-01 in the treatment of relapsed/refractory of B-cell malignancies. | From ZZSW-01 infusion to the end of the treatment at 96 weeks.
  Tumor response after ZZSW-01 infusion will be assessed according to the Lugano 2014 criteria or the 2017 ELN criteria. The Stable Disease (SD) rate will be determined.
Progressive Disease (PD) Rate of administering ZZSW-01 in the treatment of relapsed/refractory of B-cell malignancies. | From ZZSW-01 infusion to the end of the treatment at 96 weeks.
  Tumor response after ZZSW-01 infusion will be assessed according to the Lugano 2014 criteria or the 2017 ELN criteria. The Progressive Disease (PD) rate will be determined.
Objective response rate (ORR) of administering ZZSW-01 in the treatment of relapsed/refractory of B-cell malignancies. | From ZZSW-01 infusion to the end of the treatment at 96 weeks
  Objective response rate (ORR) after ZZSW-01 infusion will be evaluated according to the Lugano 2014 criteria or the 2017 ELN criteria.
Overall survival (OS) of administering ZZSW-01 in the treatment of relapsed/refractory of B-cell malignancies. | From ZZSW-01 infusion to the end of the treatment at 96 weeks
  Overall survival (OS) after ZZSW-01 infusion will be evaluated according to the Lugano 2014 criteria or the 2017 ELN criteria.
Progression-free survival (PFS) of administering ZZSW-01 in the treatment of relapsed/refractory of B-cell malignancies. | From ZZSW-01 infusion to the end of the treatment at 96 weeks
  Progression-free survival (PFS) after ZZSW-01 infusion will be evaluated according to the Lugano 2014 criteria or the 2017 ELN criteria.
Time to response (TTR) of administering ZZSW-01 in the treatment of relapsed/refractory of B-cell malignancies. | From ZZSW-01 infusion to the end of the treatment at 96 weeks
  Time to response (TTR) after ZZSW-01 infusion will be evaluated according to the Lugano 2014 criteria or the 2017 ELN criteria.
Duration of response (DOR) of administering ZZSW-01 in the treatment of relapsed/refractory of B-cell malignancies. | From ZZSW-01 infusion to the end of the treatment at 96 weeks
  Duration of response (DOR) after ZZSW-01 infusion will be evaluated according to the Lugano 2014 criteria or the 2017 ELN criteria.
Peak Level (Cmax) of CAR-T Cells | Baseline, DAY1, Day 4, Day 7, Day 14, Day 21, Day 28, Week 8, Week 12, Week 24, Week 36, Week48 or withdrawal from the study, whichever came first.
  PK parameters: The peak level (Cmax) of CAR-T cells in the peripheral blood will be measured and reported.
Pharmacodynamic (PD) characteristics of ZZSW-01 in patients with relapsed/refractory B cell malignancies | Baseline, DAY1, Day 4, Day 7, Day 14, Day 21, Day 28, Week 8, Week 12, Week 24, Week 36, Week48 or withdrawal from the study, whichever came first.
  PD parameters: including lymphocyte subgroups, CD19 positive B cell and other cell proportions, various cytokines, immunoglobulins, etc.
Time to Peak Level (Tmax) of CAR-T Cells | Baseline, DAY1, Day 4, Day 7, Day 14, Day 21, Day 28, Week 8, Week 12, Week 24, Week 36, Week48 or withdrawal from the study, whichever came first.
  PK parameters: The time to reach the peak level (Tmax) of CAR-T cells in the peripheral blood will be determined.
Area Under the Curve (AUC0-28d) of CAR-T Cells | Baseline, DAY1, Day 4, Day 7, Day 14, Day 21, Day 28, Week 8, Week 12, Week 24, Week 36, Week48 or withdrawal from the study, whichever came first.
  PK parameters: The area under the concentration-time curve from time zero to 28 days (AUC0-28d) for CAR-T cells in the peripheral blood will be calculated.
Duration of Persistence of CAR-T Cells | Baseline, DAY1, Day 4, Day 7, Day 14, Day 21, Day 28, Week 8, Week 12, Week 24, Week 36, Week48 or withdrawal from the study, whichever came first.
  PK parameters: The duration for which CAR-T cells persist in the peripheral blood will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, Ph.D&M.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: No